CLINICAL TRIAL: NCT02858167
Title: Creation of a Normal Database for FluoroDeoxyGlucose-Positron Emission Tomography (FDG-PET) Neurological Examinations: Study of Principal Inter-individual Variation Factors
Brief Title: Creation of a Normal Database for FluoroDeoxyGlucose-Positron Emission Tomography (FDG-PET) Neurological Examinations
Acronym: BDD TEP FDG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2008-A00763-52
Record Dates: First submitted 2016-07-29; First posted 2016-08-08 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FDG-PET (Experimental)
  Interventions: Device: FDG-PET

INTERVENTIONS:
Device: FDG-PET — FDG injection followed by cerebral examination with X ray spiral CT after 40 minutes and FDG-PET after 60 minutes

SUMMARY:
The purpose of this study is to define a reference population for FDG-PET neurological examinations starting from patients having FDG-PET to supervise a non-complicated lymphoma (tumor in remission, low disabling chronic tumor).

DETAILED DESCRIPTION:
This study will also check normality of cerebral functions in this population and analyse the influence of various variation factors, such as age, sex ratio, education level, professional activity and neuropsychological test results on normal data.

This database could be later used as comparison to patient images defining the gravity and localization of their cerebral functional disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patient with tumor in remission or low disabling chronic tumor
* No parenteral chemotherapy for at least 1 month
* No glucocorticoid treatment
* No general health modification (asthenia, anorexia, weight reduction)

Exclusion Criteria:

* Patient having a known neurodegenerative disorder, a general disease or physical problems that can interfere with cognitive function
* Patient with cerebral pathology history (epilepsy, vascular event, cerebral vascular malformation, tumor, severe cranial trauma, meningitis or infectious or inflammatory encephalitis, hydrocephalus, mental retardation…)
* Patient not having at least 4 years of education
* Patient having an anxiolytic or anti-depressive treatment
* Patient refusing to participate to the study
* Patient incapable to give informed consent (guardianship)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-02; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Absence of neurological impairment detected during standard neurological examination | Day 0
Mini-mental state score | Day 0
Frontal Assessment Battery score | Day 0
Mini International Neuropsychiatric Interview (DSM-IV) score | Day 0
Montgomery-Åsberg depression rating scale | Day 0
Absence of cerebral abnormalities detected with PET | Day 0
Absence of cerebral abnormalities detected with X ray spiral CT | Day 0

SECONDARY OUTCOMES:
Instrumental Activities of Daily Living evaluation | Day 0
  Evaluation of the normality of cerebral function in study population
Cerebral FDG distribution | Day 0
  Voxel-based analysis with SPM software of PET data
FDG mean activity in cerebral sections | Day 0
  Automatic measurement of FDG mean fixation in cerebral sections with NeurogamTM (Segami) software in PET data

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Laurens, Principal Investigator — Service de Médecine Nucléaire, Hôpital Central, Nancy, France; Pierre-Yves MARIE, Principal Investigator — Service de Médecine Nucléaire, Hôpital Central, Nancy, France
Locations (1):
- Service de Médecine Nucléaire, Hôpital Central, Nancy, France

IPD SHARING:
Plan to Share IPD: No